CLINICAL TRIAL: NCT03246295
Title: Identification of Gestational Diabetes Mellitus Related Urinary Biomarkers Along Pregnancy (From Early Pregnancy to Postpartum) by Using Proteomics and Metabolomics Analysis
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, wuxueyan, professor，MD, Peking Union Medical College Hospital
Other Study IDs: ZS976
Record Dates: First submitted 2017-07-23; First posted 2017-08-11 (Actual); Last update posted 2017-08-11 (Actual); Status verified 2017-08

CONDITIONS: Gestational Diabetes Mellitus
Keywords: Proteomics; Metabolomics
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urinary samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Gestational diabetes mellitus: Those women were diagnosed as gestational diabetes mellitus
  Interventions: Other: lifestyle intervention or insulin treatment
- Control: Those women were diagnosed without gestational diabetes mellitus

INTERVENTIONS:
Other: lifestyle intervention or insulin treatment — Firstly，the gestational diabetes mellitus（GDM） women were treated with lifestyle intervention.Those women were treated with insulin if their blood glucose was not well Controled.
  Groups: Gestational diabetes mellitus

SUMMARY:
Gestational diabetes mellitus (GDM) has many adverse effects on pregnant women and fetuses. At present, no prediction marker for GDM in early pregnancy is accepted. There is still a lack of recognized early predictors. This study was designed to identity valuable biomarkers for GDM.This was a prospective observed cohort study. 140 pregnant women were recruited in early pregnancy, and followed up to 6 weeks postpartum. Glucose challenge test and 75g oral glucose tolerance test were performed after 24 weeks of pregnancy, and GDM was diagnosed according to the latest ADA standard. Urinary samples were collected in the first (<12 weeks), second (24~28 weeks) and third (32~weeks) trimester of pregnancy. Urinary proteomics and metabolomics were analyzed by ultra-performance liquid chromatography tandem mass spectrometry. 15 cases of GDM women and 50 cases of control women were used for longitudinal analysis; 15 cases of GDM women and 15 cases of age matched control women were used for difference analysis.

ELIGIBILITY:
Inclusion Criteria:

-Pregnant women （<12 weeks）

Exclusion Criteria:

* with renal dysfunction
* urine routine examination abnormalities for twice
* history of urinary and reproductive system diseases
* with other chronic diseases

Ages: 18 Years to 45 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes — Pregnant women
Study Population: Pregnant women were recruited in early pregnancy, and followed up to 6 weeks postpartum
Sampling Method: Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2015-10-20 (Actual); Primary Completion 2017-09-01 (Estimated); Study Completion 2017-10-01 (Estimated)

PRIMARY OUTCOMES:
Urinary samples were analyzed | in the first (<12 weeks) trimester of pregnancy
  Urinary samples were collected and urinary proteomics and metabolomics were analyzed by ultra-performance liquid chromatography tandem mass spectrometry.

SECONDARY OUTCOMES:
Urinary samples were analyzed | in the second (24-28 weeks) trimester of pregnancy
  Urinary samples were collected and urinary proteomics and metabolomics were analyzed by ultra-performance liquid chromatography tandem mass spectrometry.
Urinary samples were analyzed | in the third (>32 weeks) trimester of pregnancy
  Urinary samples were collected and urinary proteomics and metabolomics were analyzed by ultra-performance liquid chromatography tandem mass spectrometry.

REFERENCES:
- [Derived] Duo Y, Song S, Qiao X, Zhang Y, Xu J, Zhang J, Peng Z, Chen Y, Nie X, Sun Q, Yang X, Wang A, Sun W, Fu Y, Dong Y, Lu Z, Yuan T, Zhao W. A Simplified Screening Model to Predict the Risk of Gestational Diabetes Mellitus in Pregnant Chinese Women. Diabetes Ther. 2023 Dec;14(12):2143-2157. doi: 10.1007/s13300-023-01480-8. Epub 2023 Oct 16. PMID 37843770
- [Derived] Duo Y, Song S, Zhang Y, Qiao X, Xu J, Zhang J, Peng Z, Chen Y, Nie X, Sun Q, Yang X, Wang A, Sun W, Fu Y, Dong Y, Lu Z, Yuan T, Zhao W. Relationship between serum uric acid in early pregnancy and gestational diabetes mellitus: a prospective cohort study. Endocrine. 2024 Mar;83(3):636-647. doi: 10.1007/s12020-023-03544-y. Epub 2023 Oct 2. PMID 37782356
- [Derived] Liu X, Wang X, Sun H, Guo Z, Liu X, Yuan T, Fu Y, Tang X, Li J, Sun W, Zhao W. Urinary metabolic variation analysis during pregnancy and application in Gestational Diabetes Mellitus and spontaneous abortion biomarker discovery. Sci Rep. 2019 Feb 22;9(1):2605. doi: 10.1038/s41598-019-39259-2. PMID 30796299